CLINICAL TRIAL: NCT00396071
Title: A Single-center, Double-blind, Randomized, Placebo-controlled, Cross-over Study to Assess the Effect of Vildagliptin on the Incretin Effect in Patients With Type 2 Diabetes Treated With Metformin
Brief Title: Efficacy and Safety of Vildagliptin Compared to Placebo on the Incretin Effect in Patients With Type 2 Diabetes Treated With Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2387
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin; incretin effect; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

ARMS (2):
- 1 (Experimental): Vildagliptin 100 mg qd
  Interventions: Drug: vildagliptin
- 2 (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: vildagliptin — vildagliptin 100 mg
  Other Names: Galvus
  Arms: 1
Drug: Placebo — matching placebo
  Arms: 2

SUMMARY:
This mechanistic study will evaluate the effect of vildagliptin on glucose-stimulated insulin secretion to improve the incretin effect in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes on metformin for at least 3 months and have been on a stable dose of at least 1500 mg daily for a minimum of 4 weeks
* Agreement to maintain the same dose of metformin throughout the study
* Body mass index (BMI) in the range of 22-35 kg/m2
* HbA1c in the range of 7.0 to 9.0%
* FPG <200 mg/dl (11.1 mmol/L)
* Agreement to maintain prior diet and exercise habits during the full course of the study
* Ability to comply with all study requirements and signed informed consent to participate in the study

Exclusion Criteria:

* A history of type 1 diabetes
* A history of acute metabolic diabetic complications
* Evidence of significant diabetic complications
* Insulin treatment for longer than 10 days within the past 6 months
* Treatment with any oral anti-diabetic other than metformin within 3 months prior to visit 1

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 30 Years to 78 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-10; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Change in C-peptide IAUC (0-4hr) | 2 weeks after treatment

SECONDARY OUTCOMES:
Change in insulin secretion rate (ISR) relative to glucose (0-2hr) | after 2 weeks of treatment
Change in postprandial C-peptide | after two weeks of treatment
Change in postprandial insulin | after two weeks of treatment
Change in postprandial glucagon | after two weeks of treatment
Change in postprandial GLP-1 | after 2 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Diabetes Zentrum Bad Lauterberg, Bad Lauterberg im Harz, Germany
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Result] Vardarli I, Nauck MA, Kothe LD, Deacon CF, Holst JJ, Schweizer A, Foley JE. Inhibition of DPP-4 with vildagliptin improved insulin secretion in response to oral as well as "isoglycemic" intravenous glucose without numerically changing the incretin effect in patients with type 2 diabetes. J Clin Endocrinol Metab. 2011 Apr;96(4):945-54. doi: 10.1210/jc.2010-2178. Epub 2011 Jan 14. PMID 21239518